CLINICAL TRIAL: NCT07143292
Title: A Prospective, Randomized, Parallel Trial of Famitinib Malate at Different Doses Combined With Camrelizumab for the Treatment of Recurrent and Metastatic Cervical Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Lu Huaiwu, doctor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-CervC-II-009
Record Dates: First submitted 2025-08-12; First posted 2025-08-27 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Cervical Cancer Metastatic; Cervical Cancer Recurrent
MeSH Terms: interventions — famitinib; camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): Famitinib 20 mg QD PO + Camrelizumab 200 mg IV Q3W
  Interventions: Drug: Famitinib + Camrelizumab
- Arm 2 (Experimental): Famitinib 15 mg QD PO + Camrelizumab 200 mg IV Q3W
  Interventions: Drug: Famitinib + Camrelizumab
- Arm 3 (Experimental): Famitinib 10 mg QD PO + Camrelizumab 200 mg IV Q3W
  Interventions: Drug: Famitinib + Camrelizumab

INTERVENTIONS:
Drug: Famitinib + Camrelizumab — Famitinib + Camrelizumab

SUMMARY:
This study is a prospective, randomized, parallel investigation aimed at evaluating different doses of famitinib malate (20mg, 15mg, or 10mg, once daily, respectively) by analyzing the pharmacokinetics, efficacy, safety, and tolerability of famitinib malate combined with camrelizumab at different doses. The feasibility of continuously oral administration combined with camrelizumab in reducing the incidence of adverse events (especially grade ≥3 adverse events) in patients by dose reduction while maintaining comparable efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily joined this clinical study and signed the informed consent form, demonstrating good compliance, be able to cooperate with follow-up visits;
2. Age: 18 to 75 years old (inclusive, calculated from the date of signing the informed consent);
3. Cervical cancer confirmed by histopathology, including cervical squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma;
4. It cannot be cured by surgery, radiotherapy or chemoradiotherapy;
5. Those who have received platinum-based systemic therapy for recurrent/metastatic cervical cancer; The number of previous systemic treatment lines is ≤2;
6. Has not received bevacizumab treatment in the past;
7. It can perform biopsies during the screening period and provide fresh tumor tissues for PD-L1 testing;
8. According to the RECIST v1.1 standard, the patient must have at least one measurable lesion;
9. ECOG score: 0-1 point;
10. Be able to swallow pills normally;
11. The expected survival period is ≥3 months;
12. The functions of important organs should meet the standards.

Exclusion Criteria:

1. History (within the past 5 years) or concurrent presence of other untreated malignant tumors, except for cured thyroid cancer, basal cell carcinoma, carcinoma in situ, and breast cancer that has been completely resected and has not recurred for more than 3 years;
2. Individuals who have previously received famitinib or are allergic to other monoclonal antibodies;
3. Individuals with any active, known autoimmune diseases;
4. Participants who have received systemic treatment with corticosteroids (prednisone or other equivalent hormones at a dose >10 mg/day) or other immunosuppressive agents within the past 4 weeks. In the absence of active autoimmune disease, inhaled or topical corticosteroids, as well as adrenal hormone replacement therapy at a dose ≤10 mg/day of prednisone equivalent, are permitted;
5. Known brain metastases or leptomeningeal metastases (excluding cases with brain metastases that have been stable for ≥4 weeks following radiotherapy or surgery);
6. Imaging studies at screening showing tumor invasion of the bladder or rectum, with an assessed risk of perforation by the investigator;
7. Spontaneous vaginal bleeding >30 ml/day within 2 weeks prior to randomization, or visible tumors in the vagina, with a risk of bleeding as assessed by the investigator;
8. Clinical symptoms of ascites or pleural effusion requiring drainage, or drainage of pleural or abdominal fluid within 2 weeks prior to randomization; excluding cases with imaging showing minimal ascites or pleural effusion without clinical symptoms;
9. History or current presence of idiopathic pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation-induced pulmonary inflammation (only radiologically demonstrated, those not requiring steroid treatment may be enrolled), drug-induced pneumonia, or active pneumonia during the screening period that the investigator determines precludes enrollment;
10. Uncontrolled cardiac symptoms or conditions, such as: (1) NYHA Class 2 or higher heart failure; (2) unstable angina; (3) acute myocardial infarction within the past year; (4) clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention;
11. Hypertension that is uncontrolled despite antihypertensive medication (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg);
12. Urinalysis indicating urine protein ≥2+, or quantitative urine protein testing confirming 24-hour urine protein quantification ≥1.0 g;
13. Currently receiving thrombolytic/anticoagulant therapy, with prophylactic use of low-dose aspirin (≤100 mg/day) or low-molecular-weight heparin (≤40 mg/day);
14. Patients who experienced any severe bleeding event of grade 2 or higher according to the CTCAE v5.0 criteria within 4 weeks prior to randomization;
15. Patients with imaging evidence of tumor invasion into major vessels or those deemed by the investigator to have a high likelihood of tumor invasion into major vessels during treatment, potentially leading to life-threatening hemorrhage;
16. Patients who have experienced intestinal obstruction or required parenteral nutrition within 1 month prior to randomization;
17. Patients who have experienced arterial or venous thromboembolic events within 6 months prior to randomization, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism, excluding lower extremity intermuscular venous thrombosis that, after assessment, does not require anticoagulant therapy, or thrombosis caused by catheter placement that has resolved and does not require medication;
18. Known hereditary or acquired bleeding and thrombotic tendencies (such as hemophilia, coagulation disorders, etc.);
19. Patients with radiation enteritis accompanied by bleeding symptoms, or those judged by the investigator to have a risk of risk of gastrointestinal perforation or bleeding;
20. Patients who have undergone prior radiotherapy, chemotherapy, or tumor surgery, with less than 4 weeks elapsed from the completion of treatment (last dose) to randomization (for patients with bone metastasis, palliative radiotherapy to an area <5% of the bone marrow region may be permitted up to 2 weeks prior to randomization); or patients who have taken oral molecularly targeted drugs within 5 drug half-lives prior to randomization; or adverse reactions (excluding alopecia) that have not recovered to ≤ CTCAE v5.0 Grade 1;
21. Subjects with active infections, or unexplained fever ≥ 38.5°C within 7 days prior to randomization, or those who have used antibiotics within 7 days prior to randomization;
22. Subjects with congenital or acquired immune deficiencies (e.g., HIV-infected individuals); or active hepatitis (HBV reference: HBsAg positive and HBV DNA ≥ 500 IU/mL or 1000 copies/mL; for hepatitis C: HCV antibody positive and HCV RNA > upper limit of normal);
23. Received a live vaccine within the previous 4 weeks or may receive one during the study period;
24. The investigator determines that the subject has other factors that may lead to the study being terminated prematurely, such as severe concomitant diseases (e.g., severe diabetes, spinal cord compression, superior vena cava syndrome, mental illness), severe laboratory abnormalities, or family or social factors that may affect the subject's safety or the collection of data and samples;
25. Severe non-healing wounds, ulcers, or fractures, or abdominal fistula, gastrointestinal perforation, or abdominal abscess within 6 months prior to randomization.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
progression free survival | up to approximately 2 years
  PFS is defined as from the time of randomization until the date of first documented progression or date of death from any cause, whichever came first

SECONDARY OUTCOMES:
objective response rate per RECIST v1.1 by investigator | up to approximately 2 years
  defined as the number of subjects with a best overall response (BOR) of CR (Disappearance of all target lesions) or PR (At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) divided by the number of measurable subjects with target lesion at baseline according to RECIST 1.1 criteria.